CLINICAL TRIAL: NCT07310446
Title: Collection of Samples From the United States Population for Optimization and Evaluation of Colorectal Cancer (CRC) Plasma Circulating Free-DNA (cfDNA) Marker Panel Performance (PROVE)
Brief Title: Collection of Samples From the United States Population for Optimization and Evaluation of Colorectal Cancer (CRC) Plasma Circulating Free-DNA (cfDNA) Marker Panel Performance
Acronym: PROVE
Status: Recruiting | Type: Observational
Sponsor: Universal Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CRC-US-002
Record Dates: First submitted 2025-12-01; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: colorectal; screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Patients newly diagnosed with CRC who have not yet had treatment or surgery.
- Arm B: People at average risk of CRC undergoing screening for colorectal cancer with colonoscopy.

SUMMARY:
This study is designed to prospectively collect blood samples and clinical data from patients that have been newly diagnosed with colorectal cancer and scheduled for resection surgery but are pre cancer treatment, subjects who are NOT scheduled for surgery but have histological confirmation of CRC from the diagnostic colonoscopy and clinical staging (cTMN) is available and are pr e- treatment, and patients who are at average risk of colorectal cancer and who are scheduled for routine colonoscopy examinations.

DETAILED DESCRIPTION:
The Sponsor has identified cfDNA (circulating free-DNA) alterations (including methylation, fragmentation, and copy-number variance) that allow specific detection of colorectal cancer (CRC) advanced precancerous lesions (APL) and is in the process of developing a bloodbased test for early detection of colorectal cancer. The Sponsor is performing the current study to evaluate and optimize the performance of a preliminary panel of markers to finalize the assay for the use for US population. This study is designed to prospectively collect blood samples and clinical data from patients that have been newly diagnosed with colorectal cancer and scheduled for resection surgery but are pre cancer treatment, subjects who are NOT scheduled for surgery but have histological confirmation of CRC from the diagnostic colonoscopy and clinical staging (cTMN) is available and are pre- treatment, and patients who are at average risk of colorectal cancer and who are scheduled for routine colonoscopy examinations.

ELIGIBILITY:
Inclusion Criteria:

* Arm A: Diagnosed with CRC
* Arm B: Undergoing screening with colonoscopy for CRC

Exclusion Criteria:

* Arm A: Undergoing treatment for CRC,
* Arm B: Past history of CRC

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prevalent colorectal cancer and people undergoing screening for colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 6500 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Development of assay | Baseline
  The primary objective of this study is to optimize and evaluate the performance, including sensitivity and specificity, of the preliminary cfDNA marker panel to detect CRC and APL.

SECONDARY OUTCOMES:
ML Training | Through study completion to extend up to 24 months post LPI
  A portion of the samples will be used to train the ML algorithms and for assay development activities. Another purpose of the study is to collect samples to be used in Analytical Validation (Assay Verification) and system validation.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology and Internal Medicine Specialists, Lake Barrington, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Company IP.